CLINICAL TRIAL: NCT03118960
Title: Effectiveness of the Freedom Bed and Alternating Pressure Mattress in Treatment of Pressure Injuries in Persons With Limited Mobility Due to Traumatic Brain Injury and /or Spinal Cord Injury
Brief Title: Effectiveness of the Freedom Bed as Compared to Alternating Pressure Mattress in Treatment of Pressure Injuries in Persons With Limited Mobility Due to Traumatic Brain Injury and /or Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northeast Center for Rehabilitation and Brain Injury (Other)
Collaborators: Probed Medical USA (Unknown)
Responsible Party: Principal Investigator, Annmarie Belfiglio, Occupational Therapy Coordinator, Northeast Center for Rehabilitation and Brain Injury
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Protocol 1
Record Dates: First submitted 2016-11-17; First posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Freedom Bed (Active Comparator): Bed turns and positions subjects automatically for the healing and prevention of pressure injury
  Interventions: Device: Freedom Bed
- Group II Low Air Loss/Alternating Pressure Mattress (Active Comparator): Bed provides subjects with alternating pressure with low air loss mattress for the healing and prevention of pressure injury
  Interventions: Device: Group II Low Air Loss/Alternating Pressure Mattress

INTERVENTIONS:
Device: Freedom Bed — This is an automatic rotational system in a bed designed to disburse capillary pressure
  Arms: Freedom Bed
Device: Group II Low Air Loss/Alternating Pressure Mattress — Subjects placed on the Group II Low Air Loss/Alternating Pressure Mattresses will require manual repositioning every 2 hours
  Arms: Group II Low Air Loss/Alternating Pressure Mattress

SUMMARY:
This non-randomized clinical study will compare pressure injuries and the change in pressure injuries for subjects who are placed on the Freedom Bed compared to those placed on a standard Group II Low Air Loss/Alternating Pressure Mattress in the Ventilator Unit at Northeast Center for Rehabilitation and Brain Injury. Additionally, the incidence of pneumonia, urinary tract infections, circulatory performance, sleep deprivation and caregiver self-perception on performance will be monitored and documented.

DETAILED DESCRIPTION:
Detailed Description: This study will include 9 ventilator or oxygen dependent subjects with comparable diagnoses, nutritional levels and Stage III and/or IV pressure injuries. Of the subjects selected, 5 subjects will be placed on Freedom Beds and 4 will be placed on Group II Low Air Loss/Alternating Pressure Mattresses for a period not less than 6 months. A waiver of informed consent is required prior to bed placement and data collection. Consented subjects will have primary and secondary diagnosis recorded, pressure injuries photographed and classified, assessment of ventilator/oxygen support measured, oxygenation levels, nutrition levels, and estimated cardiac condition. Subjects will receive daily treatment and wound care as prescribed by the attending physician with weekly measurements and reporting of values. Subjects will continue until they reach one of the study endpoints: 1) discharge from the ventilator unit, or 2) withdrawal of informed consent, or 3) completion of the 6-month study.

Subjects placed on Freedom Beds will be automatically turned in accordance with positions determined optimal and approved by the attending physician. All programmable turning angles, dwell times, head and leg elevations must be "dialed in" within a week of the study beginning. Any modification to the program during the study must be approved by the care team and documented accordingly.

Subjects placed on Group II Low Air Loss/Alternating Pressure Mattresses will require manual repositioning every 2 hours. All turning and/or repositioning must be timed and documented.

The primary and secondary outcome measures documented on each subject throughout the week will be collected by the Clinical Research Coordinator (CRC) on a weekly basis and submitted to the Principal Investigator. The weekly reports will then be consolidated by the CRC into a monthly report and submitted to the Institutional Review Board (IRB), Principal Investigators (PI) and Supervising Authorities (SA) for review.

ELIGIBILITY:
Inclusion Criteria:

* Subjects or their legal representative able to provide written consent for study.
* subjects must be within the height and weight limits of the beds(height range 4'2"-6' 6" , weight range 50-300 lbs.)
* subjects must have an existing treatable stage 2 or Stage 3 wound.

Exclusion Criteria:

* Subjects with unstable spinal fractures.
* Subjects with significant involuntary spasms.
* Subjects with severe scoliosis. A user must be able to lie in a partial back lying position.
* Subjects considered obese.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Pressure Ulcers | 12 Months
  Comparison between groups - Using scale for Healing (PUSH) Tool, Standardized Assessment of Pressure Injury

SECONDARY OUTCOMES:
Incidence of pneumonia in each group | 12 months
  Comparison between groups - in-house diagnosis of Pneumonia during study period by MD or sent to ER

CONTACTS AND LOCATIONS:
Locations (1):
- Northeast Center for Rehabilitation and Brain Injury, Lake Katrine, New York, United States

IPD SHARING:
Plan to Share IPD: No